CLINICAL TRIAL: NCT06454201
Title: the First Affiliated Hospital of Nanchang University
Brief Title: Robotic Natural Orifice Specimen Extraction Surgery Compared to Robotic Assisted Surgery for Median Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanchang University (Other)
Responsible Party: Principal Investigator, Taiyuan Li, professor, Nanchang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIT2024013
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-06

CONDITIONS: Natural Orifice Specimen Extraction Surgery; Middle Rectal Cancer; Robotic; Short-term Outcomes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- robotic natural orifice specimen extraction surgery for middle rectal cancer (Active Comparator): After the body is free, the tumor segment of the bowel is pulled out through the anus. Excise the tumor segment of the colon outside the anus.
  Interventions: Procedure: robotic natural orifice specimen extraction surgery
- robotic transabdominal specimen extraction surgery for middle rectal cancer (Sham Comparator): After internal mobilization, the tumor segment of the bowel was removed through an abdominal incision. Excise the tumor segment of the bowel outside the incision.
  Interventions: Procedure: robotic transabdominal specimen extraction surgery

INTERVENTIONS:
Procedure: robotic natural orifice specimen extraction surgery — After the rectum and its mesorectum were dissociated, the rectum was transected at 2 cm below the tumor by using a linear stapler. Then the rectal stump was incised and disinfected with iodophor, the protective sleeve was placed into the abdominal cavity through the assistant hole. An assistant delivered oval forceps into the pelvic cavity through the anus and used oval forceps to grip one end of the protective sleeve. Then slowly pulled out the protective sleeve. Eventually, one end of the protective sleeve was placed inside the abdominal cavity and the other outside the anus, completely covering the rectal stump and the perianal area. Tumor was pulled out of the rectal stump, then the colon was then disconnected at 10 cm above the tumor. The anvil was placed into the stump of the sigmoid colon and disinfected with iodophor, and then the anvil was delivered into the abdominal cavity. Place a circular stapler through the anus for end-to-end anastomosis of the rectum and sigmoid colon.
  Arms: robotic natural orifice specimen extraction surgery for middle rectal cancer
Procedure: robotic transabdominal specimen extraction surgery — After the rectum and its mesorectum were dissociated, the rectum was transected at 2 cm below the tumor by using a linear stapler. Take a 6cm incision through the rectus abdominis muscle in the lower left abdomen and place an incision protective cover. Cut off the intestinal tube 10cm from the upper edge of the tumor and place a stapler base. The rectal stump was sutured with purse-string suture. Place a circular stapler through the anus for end-to-end anastomosis of the rectum and sigmoid colon. After completion of digestive tract reconstruction. The pelvic and abdominal cavities were washed repeatedly with normal saline until there were no blood remained. Close the abdominal cavity layer by layer.
  Arms: robotic transabdominal specimen extraction surgery for middle rectal cancer

SUMMARY:
The purpose of this study is to evaluate the short-term outcomes of roboric natural orifice specimen extraction surgery (NOSES-II) compared to conventional assisted robotic surgery in the treatment of median rectal cancer. The main question it aims to answer is: is it safe and feasible to perform roboric natural orifice specimen extraction surgery (NOSES-II) for median rectal cancer? What are the advantages of roboric natural orifice specimen extraction surgery (NOSES-II) compared to conventional assisted robotic surgery for median rectal cancer.

DETAILED DESCRIPTION:
A major concern to the safety of the public's health is the prevalence of colorectal cancer, which is the third most prevalent cancer and has a very high fatality rate. There are multiple treatments for rectal cancer, and surgery remains one of the most important ways. Laparoscopic surgery as a minimally invasive technique for the treatment of colorectal has been confirmed by many studies to ensure its safety and reliability. Laparoscopic surgery has also been widely used in clinical. So far, NOSES, as an emerging minimally invasive technology, has caused heated discussions in the minimally invasive surgical community, especially in rectal surgery, the emergence of NOSES, which solves the problems caused by incisions in traditional surgery, improves the mental health of patients, and has good short-term efficacy. In recent years, the popularity of robotic colorectal cancer surgery has been rising, and the concepts of radical treatment, precision, and minimally invasive have been continuously refined, and NOSES surgery, as an emerging minimally invasive technology, has further reduced the impact of surgical trauma on the body, eliminated abdominal scar incision, and avoided complications related to abdominal wall incision, and has been widely used and carried out. In addition to the benefits of patients, the high-definition lens of the robotic surgery system and the flexible robotic arm greatly remove the trembling of the operator's hand, improve the flexibility and accuracy of the operator's operation, and are more conducive to challenging operations in narrow spaces. Compared with laparoscopy, the robotic surgical system has great advantages in some aspects, such as postoperative patient urination function, sexual function, surgical complications. Robotic surgical systems, combined with NOSES, may bring greater benefits to patients.

ELIGIBILITY:
Inclusion Criteria:

1. The age is more than 18 years old and less than or equal to 85 years old
2. Eastern Cooperative Oncology Group score ≤2
3. Preoperative pathological diagnosis of rectal adenocarcinoma
4. cT1-3NxM0 median rectal cancer defined by preoperative contrast-enhanced MRI
5. The maximum diameter of tumor ≤5cm on preoperative enhanced MRI
6. The body can tolerate the operation and sign the informed consent

Exclusion Criteria:

1. multiple primary colorectal cancer
2. recurrent rectal cancer
3. preoperative neoadjuvant chemoradiotherapy
4. complicated with intestinal obstruction or intestinal bleeding requiring emergency surgery
5. previous anal surgery history
6. BMI≥30kg/m2
7. severe mental illness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
The rate of all complications | 1 months after surgery
  incidence rate
The rate of all complications (Clavien-Dindo grade ≥ III ) | 1 months after surgery
  incidence rate
The rate of anastomotic complications | 1 months after surgery
  Anastomotic leakage and anastomotic bleeding

SECONDARY OUTCOMES:
operative time | Intraoperative
  minutes
estimation of blood loss | Intraoperative
  milliliters
postoperative hospital stay | 1 day after operation
  days
visual analogue pain score | 1 weeks after surgery
  score

CONTACTS AND LOCATIONS:
Overall Officials: shanping Ye, Study Chair — The First Affiliated Hospital of Nanchang University
Locations (1):
- the First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No